CLINICAL TRIAL: NCT03073824
Title: An Open-label Long-term Evaluation of a Novel Intravaginal Device in Female Patients Experiencing Sexual and Bladder Function Issues
Brief Title: A Long-term Evaluation of a Novel Intravaginal Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joylux, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JOY 1515-03
Record Dates: First submitted 2017-02-24; First posted 2017-03-08 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Pelvic Floor Disorders; Sexual Dysfunction; Stress Incontinence
MeSH Terms: conditions — Pelvic Floor Disorders; Sexual Dysfunction, Physiological; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vSculpt, model #VS1100 (Experimental): A novel intravaginal device for females
  Interventions: Device: vSculpt

INTERVENTIONS:
Device: vSculpt — Pelvic Floor Toning and Vaginal Rejuvenation Device

SUMMARY:
An open-label long-term evaluation of a novel intravaginal device in female patients experiencing sexual and bladder function issues.

DETAILED DESCRIPTION:
To determine the long-term clinical efficacy of the vSculpt therapy on treating the pelvic floor area and vaginal tissue for females who experience bladder and sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* All study participants are required to be biological females (genotype XX) to participate
* Female participants will be of adult age, over 18
* Female participants with self-reported concerns with bladder and sexual function
* Female participants who have reliable and consistent computer and internet access on a daily basis

Exclusion Criteria:

* Female participants shall not have an active sexually transmitted disease and/or infection
* Female participants who are actively undergoing chemotherapy or radiation
* Female participants who are currently taking any cancer-related or photosensitivity drugs
* Female participants who are pregnant, who may think they are pregnant, and/or actively trying to get pregnant during the clinical study

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Improvement in Patient Quality of Life as Measured by Female Sexual Response Index | 365 days
  Improvement in patient quality of life as measured by an improvement in Female Sexual Function Index (FSFI) scores.
Improvement in patient quality of life as measured by the Female Sexual Distress | 365 days
  Improvement in patient quality of life as measured by an improvement Female Sexual Distress Score (FSDS) scores.
Improvement in patient quality of life as measured by the Urogenital Distress Inventory, Short Form (UDI-6) | 365 days
  Improvement in patient quality of life as measured by an improvement Urogenital Distress Inventory, Short Form (UDI-6) scores.
Improvement in patient quality of life as measured by the Incontinence Impact Questionnaire, Short Form (IIQ-7) | 365 days
  Improvement in patient quality of life as measured by an improvement Incontinence Impact Questionnaire, Short Form (IIQ-7) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah De La Torre, MD, Principal Investigator — Seattle OB/GYN Group
Locations (2):
- United States (2):
  - Egrari Non Invasive Center, Bellevue, Washington
  - Seattle Obstetrics and Gynecology Group, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided